CLINICAL TRIAL: NCT00473265
Title: Bone Properties in Hypoparathyroidism: Effects of PTH
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: John P. Bilezikian (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor-Investigator, John P. Bilezikian, Dorothy L. and Daniel H. Silberberg Professor of Medicine and Pharmacology, Columbia University
Organization: Columbia University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AAAA5457; R01DK069350 (NIH)
Record Dates: First submitted 2007-05-14; First posted 2007-05-15 (Estimated); Results first posted 2015-07-16 (Estimated); Last update posted 2015-07-16 (Estimated); Status verified 2015-07

CONDITIONS: Hypoparathyroidism
MeSH Terms: conditions — Hypoparathyroidism | interventions — Teriparatide; Parathyroid Hormone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- PTH(1-84) (Experimental): 100mcg of PTH1-84 every other day, every day, or every three days
  Interventions: Drug: PTH

INTERVENTIONS:
Drug: PTH
  Other Names: teriparatide; Preotact; PTH1-84; rhPTH; Natpara

SUMMARY:
Whereas much information is known about the properties of bone in primary hyperparathyroidism, a disorder of parathyroid hormone (PTH) excess, virtually nothing is known about the skeleton in hypoparathyroidism, a disorder in which PTH is absent. The purpose of this research project is to test the hypothesis that the skeleton in hypoparathyroidism is abnormal in its metabolic, densitometric, geometric, biomechanical and microarchitectural features. We will also test the hypothesis that the skeleton is dependent upon PTH for normal structure and function. Using non-invasive approaches as well as direct analysis of bone itself, the human hypoparathyroid skeleton will be thoroughly characterized. With each patient serving as his/her own control, we will determine how, to what extent, and in what ways the administration of PTH restores skeletal dynamics and structure to the hypoparathyroid skeleton. In this way, we will identify those structural and dynamic elements of the skeleton that are influenced by or dependent upon PTH. Methods to be utilized include dual energy X-ray absorptiometry, quantitative central and peripheral computed tomography, geometry and size quantification, histomorphometry by standard and microCT methods, finite element analysis, biochemical bone markers, quantitative back scattered electron imaging, and Fourier Transform Infrared Spectroscopy. This research project will extend our knowledge of the skeletal effects of PTH to its deficient range and thus complete our understanding of PTH action on bone gained by our many years of studying PTH overexpression in primary hyperparathyroidism. This investigation may also provide insight into the means by which PTH helps to restore the skeleton when it is used to treat osteoporosis.

DETAILED DESCRIPTION:
A detailed description of the methods used in this study include the following: direct analysis of bone itself. skeletal dynamics and structure such as dual energy X-ray absorptiometry, quantitative central and peripheral computed tomography, geometry and size quantification, histomorphometry by standard and microCT methods, finite element analysis, biochemical bone markers, quantitative back scattered electron imaging, and Fourier Transform Infrared Spectroscopy.

ELIGIBILITY:
Inclusion Criteria:

* Hypoparathyroidism

Exclusion Criteria:

* Bisphosphonate use

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2004-05; Primary Completion 2011-01 (Actual); Study Completion 2014-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John P Bilezikian, MD, Principal Investigator — Columbia University
Locations (1):
- Columbia University, New York, New York, United States

REFERENCES:
- [Derived] Rubin MR, Zhou H, Cusano NE, Majeed R, Omeragic B, Gomez M, Nickolas TL, Dempster DW, Bilezikian JP. The Effects of Long-term Administration of rhPTH(1-84) in Hypoparathyroidism by Bone Histomorphometry. J Bone Miner Res. 2018 Nov;33(11):1931-1939. doi: 10.1002/jbmr.3543. Epub 2018 Aug 16. PMID 29972871

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 68 subjects were enrolled from 05/12/2004 to 06/19/2014 at Columbia University Medical Center.
Pre-assignment Details: The first 6 participants in the study were randomly assigned to PTH1-84 100mcg daily, 100mcg every other day, and 100mcg every three days as a pilot project to determine the correct dosing regimen.
Groups:
- PTH1-84: participants received PTH1-84 in either 100mcg daily, every other day, or every three days based on investigators clinical judgement
Period: Overall Study
Arm/Group | PTH1-84
Started | 68
Completed | 48
Not Completed | 20
Not completed — Unrelated adverse event | 5
Not completed — Off treatment early | 15

BASELINE CHARACTERISTICS:
Population: hypoparathyroidism patients who signed Consent to participate in the study
Groups:
- PTH1-84: participants recieved PTH1-84 in either 100mcg daily, every other day, or every three days based on investigators clinical judgement
Arm/Group | PTH1-84
Number analyzed (Participants) | 68
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 66
  >=65 years | 2
Age, Continuous [Mean (Standard Deviation); unit: years] | 45 (27)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 50
  Male | 18
Region of Enrollment [Number; unit: participants]
  United States | 68

OUTCOME MEASURES:

1. Primary Outcome: Requirements for Calcium Supplementation
Description: Serum and urinary calcium levels maintained by change in requirements for calcium supplementation
Time Frame: 2 years
Population: Only the first 30 participants to complete 24 months in the study were analyzed
Measure: Mean (Standard Deviation); unit: grams per day of calcium supplementation
Arm/Group | PTH1-84
Number analyzed (Participants) | 30
grams per day of calcium supplementation
  Starting requirements | 3.03 (2.32)
  Requirements at month 24 | 1.66 (1.26)

2. Secondary Outcome: Percent Change in BMD From Baseline to 24 Months by DXA
Description: Bone Mineral Density (BMD) as measured by Dual-energy X-ray absorptiometry (DXA).
Time Frame: baseline versus 24 months
Population: Only the first 30 participants who completed 24 months of the study were analyzed
Measure: Mean (Standard Deviation); unit: percentage of change to BMD
Arm/Group | PTH1-84
Number analyzed (Participants) | 30
percentage of change to BMD
  Lumbar Spine BMD | 2.9 (4)
  Femoral Neck BMD | 0.95 (.2)
  Distal 1/3 Radius BMD | -2.4 (4)

3. Secondary Outcome: Trabecular Width
Description: Trabecular width was obtained from histomorphometric assessment of percutaneous iliac crest bone biopsy. Trabecular width is the thickness of individual pieces of the spongy bone section. The structure and microscopic organization of a small piece of biopsied pelvic bone was analyzed.
Time Frame: baseline versus two years
Population: Only 16 subjects had paired bone biopsies obtained at baseline and after 24 months of PTH(1-84) treatment.
Measure: Mean (Standard Deviation); unit: micrometers
Arm/Group | PTH1-84
Number analyzed (Participants) | 16
micrometers
  Baseline | 144 (34)
  Year 2 | 128 (34)

4. Secondary Outcome: Trabecular Number
Description: trabecular number done on histomorphometric assessment of percutaneous iliac crest bone biopsy. Trabecular number is the number of individual pieces of the spongy bone section. The structure and microscopic organization of a small piece of biopsied pelvic bone was analyzed.
Time Frame: baseline versus two years
Population: Only 16 subjects had paired bone biopsies obtained at baseline and after 24 months of PTH(1-84) treatment.
Measure: Mean (Standard Deviation); unit: mm^-1
Arm/Group | PTH1-84
Number analyzed (Participants) | 16
mm^-1
  Baseline | 1.74 (0.34)
  Year 2 | 2.07 (0.5)

5. Secondary Outcome: Cortical Porosity
Description: Cortical porosity done on histomorphometric assessment of percutaneous iliac crest bone biopsy. Cortical Porosity measures how many tiny holes there are in the solid bone section. The structure and microscopic organization of a small piece of biopsied pelvic bone was analyzed.
Time Frame: baseline versus two years
Population: Only 16 subjects had paired bone biopsies obtained at baseline and after 24 months of PTH(1-84) treatment.
Measure: Mean (Standard Deviation); unit: percentage of porosity
Arm/Group | PTH1-84
Number analyzed (Participants) | 16
percentage of porosity
  Baseline | 7.4 (3.2)
  Year 2 | 9.2 (2.4)

6. Secondary Outcome: Mineralizing Surface
Description: Mineralizing surface done on histomorphometric assessment of percutaneous iliac crest bone biopsy. Mineralizing surface measures how much of bone is getting new mineral put on it. The structure and microscopic organization of a small piece of biopsied pelvic bone was analyzed.
Time Frame: baseline versus one year
Population: Only 14 subjects had paird bone biopsies obtained at baseline and after 12 months of PTH(1-84) treatment.
Measure: Mean (Standard Deviation); unit: percentage of surface
Arm/Group | PTH1-84
Number analyzed (Participants) | 14
percentage of surface
  Baseline | 0.7 (0.6)
  Year 1 | 7.1 (6.0)

ADVERSE EVENTS:
Time Frame: earliest SAE report is 8/2/05 and latest SAE report is 6/19/09
Arm/Group | PTH1-84
Serious Adverse Events (participants affected / at risk) | 15/68
Other Adverse Events (participants affected / at risk) | 68/68
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | PTH1-84 (N=68)
Infection at bone biopsy site (Infections and infestations) | 1/63 (1) — secondary to participation in study but unrelated to study drug
Right Kidney mass (Renal and urinary disorders) | 1 (1) — unlikely to be related to study participation
Abdominal Pain (Musculoskeletal and connective tissue disorders) | 2 (3) — categorized as an SAE because it involved hospitalization. unrelated to study participation
pancreatitis, accute (Gastrointestinal disorders) | 1 (1) — not related to study participation
ampullary mass (Hepatobiliary disorders) | 1 (1) — unrelated to study participation
anemia (Blood and lymphatic system disorders) | 1 (1) — categorized as a Serious Adverse Event because it involved hospitalization. unrelated to study participation
angina (Cardiac disorders) | 1 (1) — categorized as an SAE because it involved hospitalization unlikely to be related to study participation
concussion (Nervous system disorders) | 1 (1) — concussion secondary to car accident categorized as an SAE because it involved hospitalization unrelated to study participation
damage to surgical site of recent hernia repair (Surgical and medical procedures) | 1 (1) — patient fell and damaged the surgical site of a recent hernia repair categorized as an SAE because it involved hospitalization unrelated to study participation
dehydration (Blood and lymphatic system disorders) | 1 (1) — patient hospitalized with dehydration unrelated to study participation
cyst removal (Surgical and medical procedures) | 1 (1) — unrelated to study participation
symptomatic hypocalcemia (Endocrine disorders) | 4 (9) — though hypocalcemia is an anticipated syndrome of hypoparathyroidism, this event resulted in hospitalization unrelated to study participation
pneumonia (Respiratory, thoracic and mediastinal disorders) | 2 (2) — categorized as a SAE because it involved hospitalization unrelated to study participation
laryngeal spasm (Musculoskeletal and connective tissue disorders) | 1 (1) — categorized as an SAE because it involved hospitalization unrelated to study participation
Fainted (Blood and lymphatic system disorders) | 1 (1) — Due to GERD
L Oophorectomy (Reproductive system and breast disorders) | 1 (1)
Elective Surgery (Surgical and medical procedures) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PTH1-84 (N=68)
Anxiety/Irritabilty/Stress (Psychiatric disorders) | 20 (29)
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 47 (134)
Rash (Skin and subcutaneous tissue disorders) | 5 (5) — Rash locations vary from patient to patient, areas reported were face and cheeks, arms and legs and coccyx areas.
Bruising at injection site (Skin and subcutaneous tissue disorders) | 9 (9)
Chest Pain (Respiratory, thoracic and mediastinal disorders) | 8 (8)
Cold/Flu Virus/Symptoms (Infections and infestations) | 28 (32) — This adverse event refers to patients who had experienced either cold and flu virus's or symptoms
Constipation (Gastrointestinal disorders) | 7 (8)
Decrease in Urination (Renal and urinary disorders) | 7 (7)
Depression (Psychiatric disorders) | 11 (12)
Diarrhea (Gastrointestinal disorders) | 9 (9)
Dizziness (Nervous system disorders) | 21 (24)
Fatigue (Endocrine disorders) | 23 (29)
Headache/Migraine (Nervous system disorders) | 32 (42)
Temperature Sensitivity (Endocrine disorders) | 10 (11)
Hypercalcemia (Endocrine disorders) | 5 (6)
Hypertension (Blood and lymphatic system disorders) | 8 (8)
Increased Urination (Renal and urinary disorders) | 20 (22)
Insomnia (Nervous system disorders) | 16 (17)
Musculoskeletal Irritability (Musculoskeletal and connective tissue disorders) | 41 (74)
Weight Fluctuations (Metabolism and nutrition disorders) | 14 (14)
Vomitting (Gastrointestinal disorders) | 4 (4)
Increased Thirst (Renal and urinary disorders) | 14 (14)
Gastrointestinal Pain (Gastrointestinal disorders) | 18 (23)
Nausea (Gastrointestinal disorders) | 34 (47)
Decreased Appetite (Metabolism and nutrition disorders) | 10 (10)
Confusion\Disorientation (Psychiatric disorders) | 11 (13)
Bone Fracture (Musculoskeletal and connective tissue disorders) | 6 (7)
Body Swelling (Blood and lymphatic system disorders) | 4 (6)
Difficulty Breathing (Respiratory, thoracic and mediastinal disorders) | 10 (10)
Alopecia (Skin and subcutaneous tissue disorders) | 5 (5)
Arrhythmia (Cardiac disorders) | 7 (9)
Cysts (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 10 (12)
Heartburn (Gastrointestinal disorders) | 4 (4)
Infection (Infections and infestations) | 29 (42)
Kidney Stone/Kidney Pain (Renal and urinary disorders) | 8 (9)
Opthalmological Irritability/Visual Impairment (Eye disorders) | 11 (16)
Hypocalcemic Symptoms (Endocrine disorders) | 6 (6)

LIMITATIONS AND CAVEATS:
Only 16 subjects received a bone biopsy, which is why many of the measurements were only analyzed in 16 subjects. In total, data was only analyzed for the first 30 subjects analyzed for data.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No